CLINICAL TRIAL: NCT00703352
Title: Aldosterone Antagonists in Systemic Right Ventricle: a Randomized Clinical Trial.
Brief Title: Eplerenone in Systemic Right Ventricle
Acronym: EVEDES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT: 2007-002605-53
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Transposition of Great Vessels; Atrial Switch Procedure
Keywords: Transposition of the great arteries.; Transposition of the great vessels.; Mustard.; Senning.
MeSH Terms: conditions — Transposition of Great Vessels | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Eplerenone
  Interventions: Drug: Eplerenone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Eplerenone (coated tablet) 50mg daily during 12 months.

SUMMARY:
BACKGROUND: There is no clinical evidence supporting medical treatment for the failing systemic right ventricle in patients with transposition of the great vessels with atrial switch. Cardiac magnetic resonance studies have shown a significant degree of myocardial fibrosis in right ventricles in the systemic position, which predisposes to systolic and diastolic dysfunction. Aldosterone is a widely recognized neurohormonal marker involved in the formation of myocardial fibrosis and the treatment with aldosterone antagonists has shown a decrease in ventricular mass in hypertensive patients, presumably related to reduction of myocardial fibrosis.

HYPOTHESIS: Low dose of eplerenone, a selective mineralocorticoid receptor blocker, in patients with systemic right ventricle can reduce the ventricular mass by means of a reduction in myocardial fibrosis, resulting in improved systolic function.

PATIENTS AND METHODS: Randomized, double blind, parallel clinical trial comparing eplerenone (50mg daily) with placebo.

Study population: Adult patients (>18 years) diagnosed with repaired transposition of the great arteries with atrial switch (Senning or Mustard techniques) routinely followed at a tertiary referral center.

Duration: 12 months. Outcomes: Right ventricular mass, myocardial fibrosis mass and ejection fraction assessed by cardiac magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Diagnosis of transposition of the great arteries repaired with atrial switch procedures (Mustard or Senning).
* Regular follow up at tertiary referral center.

Exclusion Criteria:

* Concomitant disease with life expectancy <1 year.
* Inclusion in heart transplant waiting list.
* Basal serum creatinine level > 1.5 mg/dl.
* Basal serum potassium level > 5.0 mmol/L.
* Intolerance to the investigational medical product.
* Treatment with spironolactone or eplerenone within the previous 6 months.
* Inability to undergo magnetic resonance imaging.
* Pregnancy or breast feeding.
* Denial of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Right ventricular mass assessed by cardiac-magnetic resonance | 1 year

SECONDARY OUTCOMES:
Right ventricular ejection fraction and myocardial fibrosis mass, assessed by cardiac magnetic resonance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dos, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari de la Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Dos L, Pujadas S, Estruch M, Mas A, Ferreira-Gonzalez I, Pijuan A, Serra R, Ordonez-Llanos J, Subirana M, Pons-Llado G, Marsal JR, Garcia-Dorado D, Casaldaliga J. Eplerenone in systemic right ventricle: double blind randomized clinical trial. The evedes study. Int J Cardiol. 2013 Oct 15;168(6):5167-73. doi: 10.1016/j.ijcard.2013.07.163. Epub 2013 Jul 25. PMID 23972966